CLINICAL TRIAL: NCT06108960
Title: Comparison of Pelvic Stabilization Exercises and Proprioceptive Neuromuscular Facilitation on Pain, Disability and Functional Leg Length in Patients With Anterior Innominate Iliosacral Dysfunction.
Brief Title: Pelvic Stabilization Exercises & (PNF) on Pain, Disability & Functional Leg Length
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0159
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Anterior Innominate Iliosacral Dysfunction
Keywords: Anterior innominate Iliosacral Dysfunction; Functional leg length; Pelvic Stabilization Exercise; Proprioceptive Neuromuscular Facilitation; Disability
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive neuromuscular facilitation (Experimental): The patients will be positioned in supine lying and then contract relax will be performed on affected side of pelvis first in D1 pattern (anterior elevation and posterior depression) 3 times with 10 sec contractions and 5 sec relaxations in 1 set. Then in D2 pattern (posterior elevation and anterior depression) 3 times with 10 sec contractions and 5 sec relaxations in 1 set. 3 set of each diagonal pattern to be performed in 1 treatment session alternatively. Treatment will be given for a period of 4 days a week for 8 weeks
  Interventions: Other: Proprioceptive neuromuscular facilitation
- Pelvic stabilization exercises (Experimental): All participants will receive training programs for the eight levels of training from static to dynamic conditions. The practiced therapy method will first taught by a physical therapist with a verbal explanation and visual aids (such as photographs) in each group. The therapist will supervise all stages of the exercise therapy to ensure the patients correctly performed the exercises. The supervised exercise intervention will be conducted 3 days a week for 8 weeks.
  Interventions: Other: Pelvic stabilization exercises

INTERVENTIONS:
Other: Proprioceptive neuromuscular facilitation — Group A (Proprioceptive neuromuscular facilitation.) will be treated with Proprioceptive neuromuscular facilitation, before applying exercise, Hot pack will be applied for 15 minutes. (8 weeks, 4 sessions per week) The patients will be positioned in supine lying and then contract relax will be performed on affected side of pelvis first in D1 pattern (anterior elevation and posterior depression) 3 times with 10 sec contractions and 5 sec relaxations in 1 set. Then in D2 pattern (posterior elevation and anterior depression) 3 times with 10 sec contractions and 5 sec relaxations in 1 set. 3 set of each diagonal pattern to be performed in 1 treatment session alternatively. Treatment will be given for a period of 4 days a week for 8 weeks
  Arms: Proprioceptive neuromuscular facilitation
Other: Pelvic stabilization exercises — Group B (Pelvic stabilization exercises) will be treated with Pelvic Stabilization Exercise, before applying exercise we will apply Hot pack for 15minutes (8 weeks, 3 sessions per week).
  All participants will receive training programs for the eight levels of training from static to dynamic conditions. The practiced therapy method will first be taught by a physical therapist with a verbal explanation and visual aids (such as photographs) in each group. The therapist will supervise all stages of the exercise therapy to ensure the patients correctly performed the exercises. The supervised exercise intervention will be conducted 3 days a week for 8 weeks.
  Arms: Pelvic stabilization exercises

SUMMARY:
The aim of the study is to compare the effects of pelvic stabilization exercises and proprioceptive neuromuscular facilitation on pain, disability and functional leg length in patients with anterior innominate iliosacral dysfunction.

DETAILED DESCRIPTION:
Illiosacral Dysfunction is accompanied by an abnormal movement of the ilium in relation to the sacrum, most commonly classified as either anterior or posterior innominate dysfunction. One of the unrecognized causes of low back and pelvic pain, as well as source of pain to proximal lower extremity is sacroiliac joint (SIJ) which arises from L5, S1 and in particular if there was an associated groin pain. There is a strong consensus on the effects of stabilization exercises in patients with chronic LBP, also some evidence for its benefits in patients with SJD. The aim of the study is to compare the effects of pelvic stabilization exercises and proprioceptive neuromuscular facilitation on pain, disability and functional leg length in patients with anterior innominate rotation dysfunction.

A total of 26 patients with Anterior innominate iliosacral dysfunction will be included in the study. Ethical approval will be taken from ethical committee of Riphah Internatinal University Lahore. Non-probability convenience sampling technique will be used to divide participants into group. Sample size is twenty-six. After taking informed consent and maintaining the confidentiality of individual participant, both groups will be treated with baseline treatment via the application of Hot pack. Group A will be treated with Proprioceptive neuromuscular facilitation and Group B will be treated with Pelvic Stabilization Exercises for eight weeks. Outcome measuring tools for pain (Numeric Pain Rating Scale), Functional Disability (Modified Oswestry low back pain disability Questionnaire) and Functional Leg length (Tape Method) will be noted pre, 4th week and post treatment. Data will be Analyzed by SPSS version 29. Descriptive statistics will be used for demographics. The normality of the data will be assessed by Shapiro-Wilk test. If the data is normally distributed parametric test i.e., T-Test will be used for inter group difference while Paired Sample T-Test will be used for intra group pre and post treatment difference. If the data is not normally distributed a nonparametric test i.e., Mann-Whitney test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patient within ages of 25 and 45 years.
* Both male and female participants will be included.
* Episode of Lumbopelvic pain within the previous 6 weeks with pain radiating till the knee and associated groin pain.
* Pain and tenderness at SIJ
* The diagnostic criteria for SJD were five clinical tests Compression, Distraction, sacral thrust, thigh thrust and Gaenslen test (patient with a minimum of 3 positive results among the 5 provocation tests)
* Positive Special test for Anterior Innominate Dysfunction (Standing flexion test, Seated flexion test, Supine to sit test and Gillet test)
* NPRS = 3 to 6

Exclusion Criteria:

* Any other medical/systemic illness relevant to lower back and lower extremity
* Previous major surgery for lower back and lower extremity
* SLR Less than 45°
* Pain radiating past the knee
* Pregnant and lactating females
* Had been diagnosed by physician with a diagnosis other than SIJD
* Receiving manual therapy for the sacroiliac joint in the past 3 month

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-08 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale NPRS | 8 week
  Change from baseline the NPRS is a self-reporting or clinician-administered measuring tool that has extreme values ranging from "no pain" to "severe pain", on either horizontal or vertical line of scale. Numeric Rating Scale (NRS-11), which is an eleven-point scale in which the end points are the extremes of no pain at all (score of 0) and the worst pain the patient has ever experienced (score of 10).
Modified Oswestry low back pain disability Questionnaire | 8 week
  Change from baseline this questionnaire has been designed to give information as to how back pain has affected the ability to manage in everyday life. It consists of total of 10 questions which are scored as follow:
  This scale consists of 10 items in the form of activities of daily living with each item scoring from 0 to 5 where 0 is no difficulty in performing that activity and 5 inability to do that activity.
Measurement of Functional Leg length: (Tape Method): | 8 week
  Change from baseline the true leg length measurement or spinomalleolar distance (acceptable validity and reliability [intraclass correlation coefficient (ICC3,3) range 0.98 - 0.99] in measuring LLD) was used to assess the leg length of the subjects. A measuring tape will then use to measure from the apex of anterior superior iliac spine (ASIS) to the distal end of the medial malleolus in each leg and recorded in millimeter (mm). The following is the classification of the level of LLD: mild (< 30 mm), moderate (30 - 60 mm) and severe (> 60 mm).

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Amjad, M.Phil, Principal Investigator — Riphah International University
Locations (1):
- Sehat Medical Complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brolinson PG, Kozar AJ, Cibor G. Sacroiliac joint dysfunction in athletes. Curr Sports Med Rep. 2003 Feb;2(1):47-56. doi: 10.1249/00149619-200302000-00009. PMID 12831676
- [Background] ASAD F, HAFEEZ S, SAEED S, RIAZ S, KHAN RR, AWAN AB. Comparison of Post Isometric Relaxation of Gluteus Maximus and Static Stretching of Hip Flexors on Pain and Functional Status in Patients with Anterior Innominate Dysfunction.
- [Background] Timm KE. Sacroiliac joint dysfunction in elite rowers. J Orthop Sports Phys Ther. 1999 May;29(5):288-93. doi: 10.2519/jospt.1999.29.5.288. PMID 10342566
- [Background] Oldreive WLJJoM, Therapy M. A critical review of the literature on tests of the sacroiliac joint. 1995;3(4):157-61.
- [Background] Vaidya A, Babu VS, Mungikar S, Dobhal SJIJHS. Comparison between muscle energy technique and Mulligan's mobilization with movement in patients with anterior innominate iliosacral dysfunction. 2019;1(9).
- [Background] Shaw J, editor The role of the sacroiliac joint as a cause of low back pain and dysfunction. The First Interdisciplinary World Congress on Low Back Pain and its Relation to the Sacroiliac Joint, San Diego, CA; 1992.
- [Background] Wallin D, Ekblom B, Grahn R, Nordenborg T. Improvement of muscle flexibility. A comparison between two techniques. Am J Sports Med. 1985 Jul-Aug;13(4):263-8. doi: 10.1177/036354658501300409. PMID 4025678
- [Background] Ribeiro S, Heggannavar A, Metgud SJIJoPT, Research. Effect of mulligans mobilization versus manipulation, along with mulligans taping in anterior innominate dysfunction-A randomized clinical trial. 2019;1(1):17.
- [Background] Akram H, Bashir MS, Zia A, Noor R, Shakeel A. Comparison of muscle energy technique and mobilization with movement to reduce pain and improve functional status in subjects with anterior innominate ilio-sacral dysfunction. J Bodyw Mov Ther. 2024 Oct;40:1336-1341. doi: 10.1016/j.jbmt.2022.11.003. Epub 2022 Dec 5. PMID 39593454
- [Background] Kumar AJN. The Effectiveness of Gluteus Maximus Activation and Kinesio Taping along with Muscle Energy Technique on Pain, Alignment and Functional Activities in Subject with Anterior Innominate Rotation Dysfunction. 2022;20(12):3650-
- [Background] Singh K, Arora L, Arora RJIJoP. Effect of proprioceptive neuromuscular facilitation (PNF) in improving sensorimotor function in patients with diabetic neuropathy affecting lower limbs. 2016:332-6.
- [Background] Kamali F, Zamanlou M, Ghanbari A, Alipour A, Bervis S. Comparison of manipulation and stabilization exercises in patients with sacroiliac joint dysfunction patients: A randomized clinical trial. J Bodyw Mov Ther. 2019 Jan;23(1):177-182. doi: 10.1016/j.jbmt.2018.01.014. Epub 2018 Jan 31. PMID 30691749
- [Background] Sharma P. Effect of Proprioceptive Neuromuscular Facilitation (PNF) in Improving Muscle Control in Patient with Sacroiliac Joint Dysfunction: A Case Report. International Journal of Recent Advances in Multidisciplinary Topics. 2021;2(3):1-4.
- [Background] Altaim SASIT, Shafique SJJoIIMCQ. Maitland's Mobilization versus Mulligan's Mobilization Technique to Treat Anterior/Posterior Innominate Dysfunctions.81.
- [Background] Kahl C, Cleland JAJPtr. Visual analogue scale, numeric pain rating scale and the McGill pain Questionnaire: an overview of psychometric properties. 2005;10(2):123-8.
- [Background] Al-Hadidi F, Bsisu I, AlRyalat SA, Al-Zu'bi B, Bsisu R, Hamdan M, Kanaan T, Yasin M, Samarah O. Association between mobile phone use and neck pain in university students: A cross-sectional study using numeric rating scale for evaluation of neck pain. PLoS One. 2019 May 20;14(5):e0217231. doi: 10.1371/journal.pone.0217231. eCollection 2019. PMID 31107910
- [Background] Bashir FJIMM. Diagnosis and manipulative therapy of sacroiliac joint disorder. 2011;33(3):115-9.
- [Background] Fritz JM, Irrgang JJ. A comparison of a modified Oswestry Low Back Pain Disability Questionnaire and the Quebec Back Pain Disability Scale. Phys Ther. 2001 Feb;81(2):776-88. doi: 10.1093/ptj/81.2.776. PMID 11175676
- [Background] Sakulsriprasert P, Vachalathiti R, Vongsirinavarat M, Kantasorn J. Cross-cultural adaptation of modified Oswestry Low Back Pain Disability Questionnaire to Thai and its reliability. J Med Assoc Thai. 2006 Oct;89(10):1694-701. PMID 17128846
- [Background] Wiangkham T, Rinrit P, Choprateep M, Thamrongthanakul R, Chidnok WJCMJ. Correlation between leg length discrepancy and asymptomatic sacroiliac joint dysfunction in young males. 2022;66(1):15-21.
- [Background] Farahmand B, Ebrahimi Takamjani E, Yazdi HR, Saeedi H, Kamali M, Bagherzadeh Cham M. A systematic review on the validity and reliability of tape measurement method in leg length discrepancy. Med J Islam Repub Iran. 2019 May 26;33:46. doi: 10.34171/mjiri.33.46. eCollection 2019. PMID 31456970
- [Background] Ehsani F, Sahebi N, Shanbehzadeh S, Arab AM, ShahAli S. Stabilization exercise affects function of transverse abdominis and pelvic floor muscles in women with postpartum lumbo-pelvic pain: a double-blinded randomized clinical trial study. Int Urogynecol J. 2020 Jan;31(1):197-204. doi: 10.1007/s00192-019-03877-1. Epub 2019 Apr 23. PMID 31016337